CLINICAL TRIAL: NCT03296072
Title: A Randomized, Examiner Blind, Crossover, in Situ Erosion Study to Investigate the Efficacy of an Experimental Dentifrice in Remineralization of Previously Softened Enamel Compared to a Placebo Dentifrice
Brief Title: In Situ Erosion Study to Investigate the Effectiveness of an Experimental Toothpaste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 208166
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2019-02-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Laboratory sample analyst will be blinded to treatment received. All study products will be overwrapped to conceal any labelling.
  The dispensing staff will not be involved in any clinical assessments or laboratory analysis during the study. Dental examiner will also be blinded to the treatment received.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Test product (Experimental): Participants will apply a full ribbon of the test product (1.5 grams [g]) containing 0.254% w/w sodium fluoride and 5% KNO3.
  Interventions: Drug: 0.254% w/w sodium fluoride and 5% KNO3
- Comparator Product (Active Comparator): Participants will apply a full ribbon of the comparator product (1.5 g orally) containing 0.454% w/w stannous fluoride.
  Interventions: Drug: 0.454% w/w stannous fluoride
- Placebo Product (Placebo Comparator): Participants will apply a full ribbon of the placebo (1.5 g orally) containing 5% KNO3.
  Interventions: Drug: 5% KNO3

INTERVENTIONS:
Drug: 0.254% w/w sodium fluoride and 5% KNO3 — Dentifrice containing 0.254% w/w sodium fluoride (1150 ppm fluoride) and 5% KNO3; plus 0.25% PVM/MA copolymer and 2.5% sodium lactate. Participants will brush it on the buccal surfaces of their natural teeth for 25 timed seconds and then swish the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants will gently rinse their mouths with 15 millilitres [mL] of tap water for 10 seconds before expectorating again.
  Arms: Test product
Drug: 0.454% w/w stannous fluoride — Dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants will brush it on the buccal surfaces of their natural teeth for 25 timed seconds and then swish the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants will gently rinse their mouths with 15 mL of tap water for 10 seconds before expectorating again.
  Arms: Comparator Product
Drug: 5% KNO3 — Fluoride free placebo dentifrice containing 5% KNO3 (0 ppm fluoride), 0.25% PVM/MA copolymer and 2.5% lactate. Participants will brush it on the buccal surfaces of their natural teeth for 25 timed seconds and then swish the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants will gently rinse their mouths with 15 mL of tap water for 10 seconds before expectorating again.
  Arms: Placebo Product

SUMMARY:
This will be a randomized, controlled, single center, single- blind, 3 period, 3 treatment, cross-over, in situ design which consists of placing pre-eroded bovine enamel specimens intra orally using a palatal appliance and testing the remineralizing performance of the experimental (dentifrice containing 0.254 Percent weight by weight [%, w/w] sodium fluoride (1150 parts per million [ppm] fluoride) and 5% KNO3 [potassium nitrate]), comparator (dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride) and placebo (Fluoride free placebo containing 5% KNO3 [0 ppm fluoride] ) dentifrices 2 and 4 hours (hrs) post treatment application, based on surface micro hardness measurements. This study will be carried out in healthy adults with a maxillary dental arch suitable for the retention of the palatal appliance.

DETAILED DESCRIPTION:
The aim of this study is to investigate the performance of an experimental dentifrice formulation in promoting enamel remineralization and inhibiting post-treatment enamel demineralization in an in situ erosion model, in comparison with a fluoride-free placebo and with a marketed competitor dentifrice product. The study will have 4 visits, 1 screening visit to assess participants eligibility and 3 treatment visits to assess product efficacy, where the treatment product will be dispensed and used under the supervision of a suitably trained study site personnel. Prior to each treatment visit, there will be a washout period of a minimum of 3 days. During this period participants will use their own dentifrice for at least one day, and a fluoride free dentifrice (provided) for two days prior to the next scheduled visit (including in the morning of the scheduled visit) to minimize any carry-over effects of the fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent.
* Male and female participants who, at the time of screening, are between the ages of 18 and 65 years, inclusive.
* Participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee. No clinically significant and relevant abnormalities in medical history or oral examination.
* Male participant able to father children and female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 5 days after the last dose of assigned treatment.
* Good oral health without lesions of the oral cavity that could interfere with the study evaluations.
* Maxillary dental arch suitable for the retention of the palatal appliance
* Unstimulated salivary flow rate of at least 0.2 mL/minute and a stimulated salivary flow rate of at least 0.8 mL/minute.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are GSK employees directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 30 days prior to screening visit.
* Participation in other studies involving investigational oral care or cosmetic products within 30 days prior to screening visit.
* Acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participant (self - reported).
* Breastfeeding female participant.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients. Unwilling or unable to comply with the lifestyle guidelines described in this protocol.
* Medication that may interfere significantly with the saliva flow in the judgment of the investigator. Should new medications that may interfere with the saliva flow be added, a second salivary flow test will be performed.
* Participant with any condition that would impact on their safety or wellbeing or affect their ability to understand and follow study procedures and requirements.
* Any sign of grossly carious lesions (active), moderate or severe periodontal conditions, or severe tooth wear. Participant presenting at screening with minor caries may continue in the study if their carious lesions are repaired prior to the first treatment visit of the study.
* Wears oral appliance or orthodontia (besides participants wearing permanent lower retainers, which are eligible).
* Recent history (within the last year) of alcohol or other substance abuse. Participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20365

REFERENCES:
- [Derived] Creeth JE, Burnett GR, Souverain A, Gomez-Pereira P, Zero DT, Lippert F, Hara AT. In situ efficacy of an experimental toothpaste on enamel rehardening and prevention of demineralisation: a randomised, controlled trial. BMC Oral Health. 2020 Apr 17;20(1):118. doi: 10.1186/s12903-020-01081-y. PMID 32303206
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=208166&attachmentIdentifier=2023405a-a4d3-4a83-81a3-646cce348c22&fileName=gsk-208166-protocol-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=208166&attachmentIdentifier=6d21b0dc-6a7f-469f-9dd7-40aeb2f0005d&fileName=gsk-208166-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in United States of America.
Pre-assignment Details: A total of 68 participates were screened, out of which 62 participants were randomized in the study and 6 participants were not randomized as all the 6 participants did not meet study criteria.
Groups:
- Test Product/Comparator Product/Placebo Product: Participants in this arm received test product (0.254% weight by weight [w/w] sodium fluoride [NaF; 1150 parts per million {ppm} fluoride] and 5% potassium nitrate [KNO3]) followed by comparator (0.454% w/w stannous fluoride [SnF2; 1100 ppm fluoride]) and placebo product (5% KNO3 [0 ppm fluoride]) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 grams [g]) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing,for a timed period of 95 seconds. After expectorating the slurry, participants gently rinsed their mouths with 15 milliliters [mL] of tap water for 10 seconds before expectorating again.
- Test Product/Placebo Product/Comparator Product: Participants in this arm received test product (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3) followed by placebo (5% KNO3 [0 ppm fluoride])and comparator product (0.454% w/w SnF2[1100 ppm fluoride]) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 g) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants gently rinsed their mouths with 15 mL of tap water for 10 seconds before expectorating again.
- Comparator Product/Test Product/Placebo Product: Participants in this arm received comparator product (0.454% w/w SnF2[1100 ppm fluoride]) followed by test (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3) and placebo product(5% KNO3 [0 ppm fluoride]) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 g) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants gently rinsed their mouths with 15 mL of tap water for 10 seconds before expectorating again.
- Comparator Product/Placebo Product/ Test Product: Participants in this arm received comparator product (0.454% w/w SnF2[1100 ppm fluoride]) followed by placebo (5% KNO3 [0 ppm fluoride])and test product (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 g) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants gently rinsed their mouths with 15 mL of tap water for 10 seconds before expectorating again.
- Placebo Product/Test Product/Comparator Product: Participants in this arm received placebo product (5% KNO3 [0 ppm fluoride]) followed by test (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3) and comparator product (0.454% w/w SnF2 [1100 ppm fluoride]) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 g) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants gently rinsed their mouths with 15 mL of tap water for 10 seconds before expectorating again.
- Placebo Product/Comparator Product/Test Product: Participants in this arm received placebo product (5% KNO3 [0 ppm fluoride]) followed by comparator (0.454% w/w SnF2[1100 ppm fluoride]) and test product (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3) in Period 1, 2 and 3 respectively. Each treatment period was separated by a wash out period of minimum 3 days (including 2 day washout period using a non-fluoride toothpaste). Participants applied a full ribbon (1.5 g) of the allocated product and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, the participants gently rinsed their mouths with 15 mL of tap water for 10 seconds before expectorating again.
Period: Treatment Period 1
Arm/Group | Test Product/Comparator Product/Placebo Product | Test Product/Placebo Product/Comparator Product | Comparator Product/Test Product/Placebo Product | Comparator Product/Placebo Product/ Test Product | Placebo Product/Test Product/Comparator Product | Placebo Product/Comparator Product/Test Product
Started | 10 | 11 | 10 | 10 | 10 | 11
Completed | 10 | 11 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treament Period 1: Wash Out Period
Arm/Group | Test Product/Comparator Product/Placebo Product | Test Product/Placebo Product/Comparator Product | Comparator Product/Test Product/Placebo Product | Comparator Product/Placebo Product/ Test Product | Placebo Product/Test Product/Comparator Product | Placebo Product/Comparator Product/Test Product
Started | 10 | 11 | 10 | 10 | 10 | 11
Completed | 10 | 11 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treament Period 2
Arm/Group | Test Product/Comparator Product/Placebo Product | Test Product/Placebo Product/Comparator Product | Comparator Product/Test Product/Placebo Product | Comparator Product/Placebo Product/ Test Product | Placebo Product/Test Product/Comparator Product | Placebo Product/Comparator Product/Test Product
Started | 10 | 11 | 10 | 10 | 10 | 11
Completed | 10 | 11 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treament Period 2: Wash Out Period
Arm/Group | Test Product/Comparator Product/Placebo Product | Test Product/Placebo Product/Comparator Product | Comparator Product/Test Product/Placebo Product | Comparator Product/Placebo Product/ Test Product | Placebo Product/Test Product/Comparator Product | Placebo Product/Comparator Product/Test Product
Started | 10 | 11 | 10 | 10 | 10 | 11
Completed | 10 | 11 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treament Period 3
Arm/Group | Test Product/Comparator Product/Placebo Product | Test Product/Placebo Product/Comparator Product | Comparator Product/Test Product/Placebo Product | Comparator Product/Placebo Product/ Test Product | Placebo Product/Test Product/Comparator Product | Placebo Product/Comparator Product/Test Product
Started | 10 | 11 | 10 | 10 | 10 | 11
Completed | 10 | 11 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
Groups:
- Overall Participants: All randomized participants were included for baseline evaluation. Participants applied a full ribbon of the test (0.254% w/w NaF [1150 ppm fluoride] and 5% KNO3), comparator (0.454% w/w SnF2[1100 ppm fluoride]) and placebo product (5% KNO3 [0 ppm fluoride]) and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth, without further brushing, for a timed period of 95 seconds. After expectorating the slurry, participants gently rinsed with 15 mL of tap water for 10 seconds before expectorating again.
Arm/Group | Overall Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 42
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: % Surface Micro Hardness Recovery (SMHR; Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to a Fluoride Free Placebo Dentifrice to Enhance Remineralization of Enamel)
Description: The %SMHR was calculated to assess the changes in mineralization status of enamel specimens. The mean indent length (micrometer) from five Knoop microindentations within each specimen was measured at baseline (B), after the first erosive challenge (E1), and after 2 and 4 hours intraoral phase (R). An increase in the indentation length compared to the baseline indicates softening of the enamel surface while decrease in the indentation length represents re-hardening of enamel surface. The %SMHR was calculated as : %SMHR = [(E1-R)/(E1-B)]*100. Greater values of %SMHR indicate that greater remineralization has occurred, thus higher values are more favorable.
Time Frame: After 4 hrs following single exposure of treatment
Population: The Intent-to-Treat (ITT) population was comprised of all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline (post-treatment) primary efficacy evaluation. This population was based on the treatment to which the participant was randomized.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMHR
Groups:
- Test Product: Participants applied a full ribbon of the test product (1.5 g) containing 0.254% w/w NaF (1150 ppm fluoride) and 5% KNO3 and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth for 95 timed seconds. After expectorating the slurry, participants gently rinsed their mouth with 15 mL of tap water for 10 seconds before expectorating again.
- Placebo Product: Participants applied a full ribbon of the placebo (1.5 g) containing 5% KNO3 (0 ppm fluoride) and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth for 95 timed seconds. After expectorating the slurry, participants gently rinsed their mouth with 15 mL of tap water for 10 seconds before expectorating again.
Arm/Group | Test Product | Placebo Product
Number analyzed (Participants) | 62 | 62
Percentage SMHR | 29.67 (1.12) | 21.98 (1.12)
Statistical Analysis 1: Comparison: Test Product vs Placebo Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 7.69, 95% CI 2-sided [5.18 to 10.19] — Difference is first-named treatment minus second-named treatment such that a positive difference favors the first named treatment

2. Secondary Outcome: % Relative Erosion Resistance (RER; Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to a Fluoride Free Placebo Dentifrice to Inhibit Demineralization of Enamel)
Description: The %RER was calculated to assess the ability of treated enamel specimens to provide a combined benefit in terms of enhanced remineralization and acid resistance of the enamel. The mean indent length (micrometer) from five Knoop microindentations within each specimen was measured at baseline (B), after the first erosive challenge (E1), and after the second erosive challenge (E2) (E2 is measured for after both 2 and 4 hours of remineralization). An increase in the indentation length compared to the baseline indicates softening of the enamel surface while decrease in the indentation length represents re-hardening of enamel surface. The %RER was calculated as : %RER = [(E1-E2)/ (E1-B)]*100. Higher values of %RER indicate greater resistance to erosion, thus higher values are more favorable.
Time Frame: After 4 hrs following single exposure of treatment
Population: The ITT population was comprised of all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline (post-treatment) primary efficacy evaluation. This population was based on the treatment to which the participant was randomized.
Measure: Least Squares Mean (Standard Error); unit: Percentage RER
Arm/Group | Test Product | Placebo Product
Number analyzed (Participants) | 62 | 62
Percentage RER | -23.65 (1.96) | -56.94 (1.96)
Statistical Analysis 1: Comparison: Test Product vs Placebo Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 33.29, 95% CI 2-sided [28.89 to 37.68] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Enamel Fluoride Uptake (EFU; Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to a Fluoride Free Placebo Dentifrice to Promote Fluoride Uptake in Enamel)
Description: The EFU was measured to determine the amount of fluoride incorporation into the model erosive lesions. Each enamel specimen drilled to a depth of approximately 100 μm using a microdrill, through the entire lesion (four cores per specimen). The enamel powder pooled from four drilling samples was then, dissolved in a known volume of perchloric acid and immediately analyzed for fluoride content using a calibrated fluoride specific electrode. The amount of fluoride-uptake by enamel was calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as microgram fluoride per square centimeter (μgF/cm^2). Higher values of EFU indicate greater incorporation of fluoride into the enamel and are thus more favorable.
Time Frame: After 4 hrs following single exposure of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Microgram fluoride per square centimeter
Arm/Group | Test Product | Placebo Product
Number analyzed (Participants) | 62 | 62
Microgram fluoride per square centimeter | 2.98 (0.09) | 1.17 (0.09)
Statistical Analysis 1: Comparison: Test Product vs Placebo Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 1.81, 95% CI 2-sided [1.59 to 2.04] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: % SMHR (Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to Comparator Containing 1100 Ppm Fluoride)
Description: The %SMHR was calculated to assess the changes in mineralization status of enamel specimens. The mean indent length (micrometer) from five Knoop microindentations within each specimen was measured at baseline (B), after the first erosive challenge (E1), and after 2 and 4 hours intraoral phase (R). An increase in the indentation length compared to the baseline indicates softening of the enamel surface while decrease in the indentation length represents re-hardening of enamel surface. The %SMHR was calculated as: %SMHR = [(E1-R)/(E1-B)]*100. Greater values of %SMHR indicate that greater remineralization has occurred, thus higher values are more favorable.
Time Frame: After 4 hrs following single exposure of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage SMHR
Groups:
- Comparator Product: Participants applied a full ribbon of the placebo (1.5 g) containing 0.454% w/w SnF2 (1100 ppm fluoride) and brushed the buccal surfaces of their natural teeth for 25 timed seconds and then swished the resulting toothpaste slurry around the mouth for 95 timed seconds. After expectorating the slurry, participants gently rinsed their mouth with 15 mL of tap water for 10 seconds before expectorating again.
Arm/Group | Test Product | Comparator Product
Number analyzed (Participants) | 62 | 62
Percentage SMHR | 29.67 (1.12) | 22.10 (1.12)
Statistical Analysis 1: Comparison: Test Product vs Comparator Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 7.57, 95% CI 2-sided [5.07 to 11.07] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: % RER (Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to Comparator Containing 1100 Ppm Fluoride)
Description: as for outcome 2
Time Frame: After 4 hrs following single exposure of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage RER
Arm/Group | Test Product | Comparator Product
Number analyzed (Participants) | 62 | 62
Percentage RER | -23.65 (1.96) | -34.63 (1.96)
Statistical Analysis 1: Comparison: Test Product vs Comparator Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 10.98, 95% CI 2-sided [6.58 to 15.37] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: EFU (Comparison of 1150 Ppm Fluoride and 5% KNO3 Dentifrice Relative to Comparator Containing 1100 Ppm Fluoride)
Description: as for outcome 3
Time Frame: After 4 hrs following single exposure of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Microgram fluoride per square centimeter
Arm/Group | Test Product | Comparator Product
Number analyzed (Participants) | 62 | 62
Microgram fluoride per square centimeter | 2.98 (0.09) | 2.01 (0.09)
Statistical Analysis 1: Comparison: Test Product vs Comparator Product; Test type: Other; p < .0001, ANOVA; From ANOVA with fixed factors for study period and treatment, and a random effect for participant; Difference of Least Square mean = 0.97, 95% CI 2-sided [0.75 to 1.20] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Test Product | Comparator Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 8/62 | 6/62 | 10/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=62) | Comparator Product (N=62) | Placebo Product (N=62)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral Mucosal Erthyema (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Bactetial Overgrowth (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sinusistis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthopod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burn Oral Cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Palate Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic Ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periodic limb movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03296072/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03296072/SAP_001.pdf